CLINICAL TRIAL: NCT02072252
Title: Mobile Phone and Internet-Based Intervention for Vulnerable Youth
Brief Title: Mobile Phone App for Depression and Anxiety in Young Men Who Are Attracted to Men
Acronym: TODAY!
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The app was not completed in time to conduct a clinical trial on it within the funding grant's award period
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michelle Burns, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00061284; K08MH094441 (NIH)
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Depressive Symptoms; Anxiety Generalized
Keywords: Depression; Anxiety; Mobile Phone; Cellular Phone; Mobile Application; Mobile Intervention; App; mHealth; eHealth; Technology Assisted; Internet; Cognitive Behavioral Therapy; LGBT; Sexual Minorities; Gay; Bisexual; Same Sex Attraction; Males; Men; Youth; Adolescents; Young Adults
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder; Anxiety Disorders; Alzheimer Disease; Homosexuality; Bisexuality; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App teaching cognitive behavioral skills (Experimental): App teaching cognitive behavioral skills. This mobile phone application ("app") teaches cognitive behavioral techniques to help participants manage their mood, for example by providing information, interactive tools and tips, and a mood tracker. A coach will support participants as they use the app via phone calls and email contacts.
  Interventions: Behavioral: Mobile Phone Application
- Wait-list with referrals (No Intervention): 10-week wait-list control condition in which participants will be provided with and encouraged to use mental health referrals to resources in the community. After the 10-week waiting period, control group participants will have the option to receive the mobile phone application and coaching.

INTERVENTIONS:
Behavioral: Mobile Phone Application — Mobile phone app teaching cognitive behavioral skills
  Other Names: TODAY!
  Arms: App teaching cognitive behavioral skills

SUMMARY:
The purpose of this study is to determine whether a mobile phone application ("app") for symptoms of depression and anxiety is practical and acceptable to young men who are attracted to men, and whether it reduces their anxiety and depressive symptoms. The investigators will also evaluate whether reductions in symptoms are maintained over a 10 week follow-up period after young men complete the mobile phone intervention.

DETAILED DESCRIPTION:
The aim of this study is to conduct a small randomized controlled trial (RCT) for a 10-week, culturally tailored mobile phone intervention that uses principles of cognitive behavioral therapy (CBT) to reduce anxiety and depression among young men who are sexually attracted to other males.

The primary purpose of the RCT is to collect feedback about the intervention from the participants. This feedback, along with usage data on which features are used more or less often by the participants, and how the features are used, will be evaluated to make improvements to the intervention. The investigators will also assess clinical outcomes (such as anxiety and depressive symptoms). Outcomes will be monitored pre-, mid-, and post-treatment, as well as twice over a 10 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male birth sex and male gender identity
* Reports sexual attraction toward males
* Is between 17-20 years of age
* Is able to speak and read English
* Resides in the Chicago metropolitan area (i.e., Chicago or suburbs of Cook County)
* Currently owns a mobile phone that is compatible with the intervention application, and believes he will be able to keep using this mobile phone for the next 10 weeks
* A score of 10 or more on the Patient Health Questionnaire-9 or 5 or more on the GAD-7

Exclusion Criteria:

* Has visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of the Internet or mobile phone
* Per self-reported history or the Mini-International Neuropsychiatric Interview, has ever been diagnosed with a psychotic disorder or bipolar disorder, or is currently diagnosed with obsessive compulsive disorder or substance dependence, or has been diagnosed in the past five years with posttraumatic stress disorder, dissociative disorder, or eating disorder; or evidences another condition that indicates this intervention may be insufficient
* Has ever been hospitalized for psychiatric reasons or attempted suicide, or has a score of 4 or more on the Columbia Suicide Severity Rating Scale, or reports non-suicidal self-injury of a nature that suggests this intervention may be insufficient
* Is participating in "Crew 450," "Keep It Up," "My Peeps," or "Q2"
* Reports currently being in Illinois Department of Child and Family Services (DCFS) custody
* Reports currently being in psychotherapy
* Initiation, discontinuation, or adjustment of antidepressant medication in the past 4 weeks
* Less than an 8th grade reading level
* Does not log into the app within 3 days of being sent the link.
* Does not have an email address

Ages: 17 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 0 (Actual)
Dates: Start 2017-08-14 (Estimated); Primary Completion 2017-08-14 (Estimated); Study Completion 2017-08-14 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | post-intervention (10 weeks)
  Self-report measure of depressive symptoms
GAD-7 | post-intervention (10 weeks)
  Self-report measure of anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Michelle N Burns, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Background] Burns MN, Montague E, Mohr DC. Initial design of culturally informed behavioral intervention technologies: developing an mHealth intervention for young sexual minority men with generalized anxiety disorder and major depression. J Med Internet Res. 2013 Dec 5;15(12):e271. doi: 10.2196/jmir.2826. PMID 24311444